CLINICAL TRIAL: NCT03190590
Title: Neurophysiological and Functional Mechanisms of Motor Control and Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17-00328
Record Dates: First submitted 2017-06-14; First posted 2017-06-19 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Transcranial Direct Current Stimulation
Keywords: transcranial magnetic stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Transcranial direct current stimulator (tDCS) (Active Comparator): tDCS is delivered noninvasively via electrodes applied to the surface of the head, and a mild electrical current is given during motor training.
  Interventions: Procedure: tDCS-NeuroConn.
- Transcranial magnetic stimulation (TMS) (Active Comparator): TMS is delivered noninvasively via a hand-held coil applied to the surface of the head, and a magnetic pulse probes cortical circuitry [this is not repetitive TMS and so does NOT modulate brain excitability.]
  Interventions: Procedure: TMS - Magstim.
- Sham-tDCS (Placebo Comparator): delivered by briefly turning on and off the stimulator at the beginning of training, which mimics the sensation of true stimulation.
  Interventions: Procedure: Sham tDCS

INTERVENTIONS:
Procedure: tDCS-NeuroConn. — tDCS is delivered noninvasively via electrodes applied to the surface of the head, and a mild electrical current is given during motor training.
  Arms: Transcranial direct current stimulator (tDCS)
Procedure: TMS - Magstim. — TMS is delivered noninvasively via a hand-held coil applied to the surface of the head, and a magnetic pulse probes cortical circuitry [this is not repetitive TMS and so does NOT modulate brain excitability
  Arms: Transcranial magnetic stimulation (TMS)
Procedure: Sham tDCS — delivered by briefly turning on and off the stimulator at the beginning of training, which mimics the sensation of true stimulation.
  Arms: Sham-tDCS

SUMMARY:
Noninvasive stimulation of the central nervous system, including transcranial magnetic stimulation (TMS) and transcranial direct current stimulation (tDCS), has been increasingly used in the investigation of cortical plasticity. The purpose of our study is to understand mechanistically-at the neurophysiological and systems levels-how the brain learns new motor skills. We propose to study the acquisition, consolidation, and retention of motor skill learning in healthy subjects. At the behavioral level, we will use movement kinematics to quantify and characterize movement, which allow us to infer functional strategies used by the brain to reduce movement errors. At a neurophysiological level, we will use TMS to document changes in cortical circuitry, which will allow us to infer neuroplastic changes possibly subserving these strategies. At a systems level, we will enhance motor system excitability using tDCS, which will enable us to infer the contribution of the stimulated area to the motor system's ability to learn new skills.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed dominance
* Ability to give informed consent

Exclusion Criteria:

* active and/or chronic neurological, psychiatric (including depression), or medical conditions
* psychoactive medication use
* active drug/alcohol dependence or abuse history
* homelessness or other social situation that would preclude consistent visits
* history of head injury (including neurosurgery)
* history of seizure
* inability to comprehend or participate in the procedures involved
* metal in the head (besides in mouth), such as implanted electrodes or devices, shrapnel, surgical clips, or fragments from welding/metalwork
* implanted devices (such as cardiac pacemakers, medical pumps, or intracardiac lines) in the thorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Motor skill gain from day 1 to day 5 | 5 Days
  defined as an improvement in performance accuracy at fixed movement speeds (see 5.2 for description of task and outcome). The delta in accuracy between day 1 and day 5 equates to motor skill learning.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Schambra-Griesemer, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States